CLINICAL TRIAL: NCT05352997
Title: Key Factors of Target Serum Concentrations Attainment From Beta-lactams Therapeutic Drug Monitoring in Critically Ill Patients
Brief Title: Beta-lactams Therapeutic Drug Monitoring in Critically Ill Patients
Acronym: SPT BETALACT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2021/HG-01
Record Dates: First submitted 2022-04-25; First posted 2022-04-29 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2022-04

CONDITIONS: Infectious Disease
Keywords: beta-lactam; lCU
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: on-target beta-lactams serum concentration: Patients with on-target beta-lactams serum concentration during 1st dosing
- Group 2: off-target beta-lactams serum concentration: Patients with off-target beta-lactams serum concentrations during 1st dosing
- Group 3: off-target beta-lactams plasma concentration:: Patients with high beta-lactams plasma concentrations during 1st dosing

SUMMARY:
The population of these monocentric and retrospective study includes patients hospitalized in one of the critical care services of Nîmes' community hospital.

The objective is to determine the key factors that lead to satisfactory beta-lactams serum concentrations in critically ill patients.

Clinical and biological features, as well as risk scores are collected and recorded into an electronic Case Report Form.

The primary outcome is to show the main characteristics related to adequate beta-lactams serum concentrations in critically ill inpatients.

Secondary outcomes include the key factors related to inadequate beta-lactams serum concentrations in critically ill inpatients, Therapeutic Drug Monitoring (TDM) impact in the achievement of target beta-lactams serum concentration and the correlation between Aminoglycosides and Beta-lactams serum concentrations. Do both antibiotics have similar elimination kinetics ?

ELIGIBILITY:
Inclusion Criteria:

* Patient aged at least (≥) 18 years of age.
* Patient (or his representative for patients unable to give their consent) has given his free and informed consent and has signed the consent form.
* Patient affiliated to the health insurance scheme
* Patient hospitalized in one of the critical care services of Nimes' community hospital with at least one beta-lactam treatment
* Patient with at least one beta-lactam TDM during his stay

Exclusion Criteria :

* Patient who did not consent the use of his personal data
* Patients under maintenance of justice, tutelage or legal guardianship
* Patient previously included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to a critical care unit and treated for an infectious episode with beta-lactam, who received a Therapeutic Drug Monitoring. All patients older than 18 years recorded between 1/1st/2018 and 3/4th/2021 were included.
Sampling Method: Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
To identify factors associated with adequate beta lactam plasma concentrations on the first sample | Day 7
  Determinants of adequate beta-lactams plasma concentrations using a univariate, then a multivariate analysis on patients 'characteristics at baseline and on the day of TDM

SECONDARY OUTCOMES:
To identify factors related with on-target beta-lactams plasma concentrations on the second sample | Day 7
  Risk factors of inadequate beta-lactam plasma concentrations using a univariate, then a multivariate analysis on patients 'characteristics at baseline and on the day of TDM.
To identify factors related with on-target beta-lactams plasma concentrations on the second sample | Day 7
  Proportion of on target 2nd dosing after inadequate first dosing
Impact of TDM | Day 7
  Mean number of TDM per patient with off-target first dosing and delay to achieve target plasma concentrations.
To assess if beta-lactams and Aminoglycosides have the same elimination kinetic | Day 7
  Linkage between beta-lactams and aminoglycosides' trough concentrations for patients concurrently treated by both antibiotics.

CONTACTS AND LOCATIONS:
Overall Officials: Claire ROGER, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gandega H, Poujol H, Mezzarobba M, Muller L, Boyer JC, Lefrant JY, Leguelinel G, Roger C. Determinants of beta-lactam PK/PD target attainment in critically ill patients: A single center retrospective study. J Crit Care. 2024 Oct;83:154828. doi: 10.1016/j.jcrc.2024.154828. Epub 2024 May 17. PMID 38759580